CLINICAL TRIAL: NCT04508114
Title: The Effectiveness of Technology-assisted Index on Improving Hand Hygiene of Registered Nurses - An Experimental Research
Brief Title: Technology-assisted Index on Improving Hand Hygiene of Registered Nurses
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 202006019RINB
Record Dates: First submitted 2020-08-05; First posted 2020-08-11 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-07

CONDITIONS: Hand Hygiene
Keywords: nurse; hand washing; ATP

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): Participants in the control group will not receive the ATP testing result (pretest) immediately until finished the research.
- experimental group (Experimental): Participants in the experimental group will be informed the ATP testing result (pretest) and receive the explanation by research assistant.
  Interventions: Behavioral: Technology-assisted Index

INTERVENTIONS:
Behavioral: Technology-assisted Index — The participant will be informed the ATP testing result and explanation in pretest.
  Arms: experimental group

SUMMARY:
In 2009, the World Health Organization (WHO) recommended the use of a multi-faceted, multi-modal hand hygiene strategy (Five Moments for Hand Hygiene) to improve hand hygiene compliance among healthcare staff. The outbreak of coronavirus disease 2019 (COVID-19) has rapidly spread globally. The novel coronavirus is characterized by rapid human-to-human transmission. Hand washing is a part of measures recommended by the World Health Organization (WHO) to avoid contracting COVID-19.The purpose of this study was to use adenosine triphosphate (ATP) testing and direct observation for improving hand hygiene and compliance in nurse.

DETAILED DESCRIPTION:
The purpose of this study was to use adenosine triphosphate (ATP) testing and direct observation as technology-assisted index on improving hand hygiene and compliance in nurse.

ELIGIBILITY:
Inclusion Criteria:

* (1)Day shift nurse on cancer ward,(2)who speak in Taiwanese and Mandarin,(3)and are willing to participate in the study.

Exclusion Criteria:

* (1)There is any wound or scar on hand.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-08-10 (Actual); Primary Completion 2022-05 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Demographics | Pre-test
  gender, age, education, nursing job tenure, job tenure in ward
Knowledge of My 5 Moments for Hand Hygiene | Pre-test
  The assessment consisted of 5 questions ,including (1)before touching a patient,(2)before clean/aseptic procedures,(3)after body fluid exposure/risk,(4)after touching a patient, (5)and after touching patient surroundings.The participant can get one point for a correct answer.Total scores range from 0 to 5.
Knowledge of My 5 Moments for Hand Hygiene (Post-test) | Immediately after completing the pre-test.
  The assessment consisted of 5 questions ,including (1)before touching a patient,(2)before clean/aseptic procedures,(3)after body fluid exposure/risk,(4)after touching a patient, (5)and after touching patient surroundings.The participant can get one point for a correct answer.Total scores range from 0 to 5.
Frequency of performing My 5 Moments for Hand Hygiene | Pre-test
  The assessment is a 5-point Likert scale with 5 items ,including (1)before touching a patient,(2)before clean/aseptic procedures,(3)after body fluid exposure/risk,(4)after touching a patient, (5)and after touching patient surroundings,from 1 to 5 that measure the frequency of performing the hand hygiene,so that higher scores indicate higher implementation of My 5 Moments for Hand Hygiene in the last week.
Frequency of performing My 5 Moments for Hand Hygiene (Post-test) | Immediately after completing the pre-test.
  The assessment is a 5-point Likert scale with 5 items ,including (1)before touching a patient,(2)before clean/aseptic procedures,(3)after body fluid exposure/risk,(4)after touching a patient, (5)and after touching patient surroundings,from 1 to 5 that measure the frequency of performing the hand hygiene,so that higher scores indicate higher belief of conducting My 5 Moments for Hand Hygiene in the next week.
Attitude on hand hygiene | Pre-test
  The assessment is a 5-point Likert scale with 1 items ,including the general attitude about the hand hygiene on working,so that higher scores indicate higher confident of hand hygiene.
Attitude on hand hygiene (Post-test) | Immediately after completing the pre-test.
  The assessment is a 5-point Likert scale with 1 items ,including the general attitude about the hand hygiene on working,so that higher scores indicate higher confident of hand hygiene.
ATP testing | Pre-test
  The 3M™ Clean-Trace™ Surface ATP test is a single-use test device that contains a swab for the collection of a sample from a surface. The swab is pre-moistened with a cationic agent to aid in the collection of soil and the release of Adenosine Tri-Phosphate (ATP) from intact cells.Upon activation of the test, reagent in the cuvette of the test device reacts with ATP collected on the swab to produce light.The intensity of the light is proportional to the amount of ATP and therefore the degree of contamination. Measurement of the light requires the use of a 3M™ Clean-Trace™ NG Luminometer and the results are displayed in Relative Light Units (RLU).ATP is an indicator of organic residues and microorganisms. Detection of ATP is used to rapidly assess the standards of hygiene and sanitation procedures for surfaces and equipment.
ATP testing (Post-test) | Immediately after completing the pre-test.
  The 3M™ Clean-Trace™ Surface ATP test is a single-use test device that contains a swab for the collection of a sample from a surface. The swab is pre-moistened with a cationic agent to aid in the collection of soil and the release of Adenosine Tri-Phosphate (ATP) from intact cells.Upon activation of the test, reagent in the cuvette of the test device reacts with ATP collected on the swab to produce light.The intensity of the light is proportional to the amount of ATP and therefore the degree of contamination. Measurement of the light requires the use of a 3M™ Clean-Trace™ NG Luminometer and the results are displayed in Relative Light Units (RLU).ATP is an indicator of organic residues and microorganisms. Detection of ATP is used to rapidly assess the standards of hygiene and sanitation procedures for surfaces and equipment.

CONTACTS AND LOCATIONS:
Overall Officials: Wei-Wen Wu, PhD, Principal Investigator — National Taiwan University, College of Medicine
Locations (1):
- NTUH, Taipei, Taiwan, 10051, Taiwan